CLINICAL TRIAL: NCT01382173
Title: Monitoring Of Helsingborg Acute Knee Injuries (MOHAK) to Understand Osteoarthritis Development After Injury.
Brief Title: Monitoring Of Helsingborg Acute Knee Injuries (MOHAK)
Status: Terminated | Type: Observational
Sponsor: Lund University (Other)
Collaborators: The Swedish Research Council (Other Government); Crafoord Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: MOHAK-11
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Knee Injury; Knee Osteoarthritis
Keywords: Knee injury; Osteoarthritis; Anterior Cruciate Ligament injury; Patellar dislocation
MeSH Terms: conditions — Knee Injuries; Osteoarthritis, Knee; Osteoarthritis; Anterior Cruciate Ligament Injuries; Patellar Dislocation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Joint fluid, Serum & Plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
Using magnetic resonance imaging (MRI), laboratory analyses and patient reported outcomes, the overall aim of this study is to investigate structural injuries and biochemical alterations in the acutely injured knee and to relate these findings to clinical outcomes at various time points.

ELIGIBILITY:
Inclusion Criteria:

1. Age 12-40 years at inclusion (inclusion of patients younger than 18 will require parental approval)
2. A history of knee injury not more than 4 weeks prior to inclusion
3. Agreement and informed consent to participate in the study

Exclusion Criteria:

1. Any MRI contra-indications (such as extreme obesity, metal implants, claustrophobia etc.)
2. Pregnancy
3. A history of deep vein thrombosis (DVT) or a disorder of the coagulative system
4. General disease that effects physical function or systemic medication/abuse of steroids
5. Any other condition or treatment interfering with the completion or assessment of the trial.

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: We will recruit approximately 150 patients annually over 3-4 years with the goal of including at least:
  * 200 knees with isolated or combined ACL injuries
  * 50 isolated meniscus tears
  * 50 primary patellar dislocations
  * 50 contusions without ligamentous, cartilage or meniscus injury.
  Patients will be recruited using two different strategies:
  1. Those seeking medical care at the orthopedic emergency room (ER) at Helsingborg hospital
  2. Those referred to the orthopedic outpatient health care unit of Helsingborg hospital due to an acute knee injury by their primary health care unit will be scheduled for a clinical visit for baseline assessment (visit 1) within four weeks from their injury. To facilitate recruitment, primary care units in the local area of Helsingborg will be offered an opportunity to refer all patients with rotational knee trauma and effusion directly to the orthopedic outpatient care unit.
Sampling Method: Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score (KOOS) | 5 yrs

SECONDARY OUTCOMES:
Radiographic osteoarthritis | 5 yrs

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Orthopedics, Helsingborg hospital, Helsingborg, Sweden